CLINICAL TRIAL: NCT02806752
Title: Multicenter Randomized Controlled Study of Intravitreal Ranibizumab and Triamcinolone Acetonide Combination Therapy Versus Ranibizumab Monotherapy in Patients With Polypoidal Choroidal Vasculopathy
Brief Title: Intravitreal Ranibizumab and TA Combination Therapy vs. Ranibizumab Monotherapy in Polypoidal Choroidal Vasculopathy
Acronym: RANTA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aier School of Ophthalmology, Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB2016006
Record Dates: First submitted 2016-04-17; First posted 2016-06-21 (Estimated); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Wet Macular Degeneration
Keywords: Polypoidal Choroidal Vasculopathy
MeSH Terms: conditions — Wet Macular Degeneration; Polypoidal Choroidal Vasculopathy | interventions — Triamcinolone Acetonide; Ranibizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ranibizumab + Triamcinolone Acetonide (Experimental): intravitreal injection: Ranibizumab 0.5mg + Triamcinolone Acetonide 2mg
  Interventions: Drug: Triamcinolone Acetonide; Drug: Ranibizumab
- Ranibizumab (Active Comparator): intravitreal injection: Ranibizumab 0.5mg
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Triamcinolone Acetonide — Intravitreal inject 0.5mg of Ranibizumab and 2mg of Triamcinolone Acetonide.
  Other Names: RANTA
  Arms: Ranibizumab + Triamcinolone Acetonide
Drug: Ranibizumab — Intravitreal inject 0.5mg of Ranibizumab.
  Other Names: RAN

SUMMARY:
The purpose of this study is to evaluate the effects and safety of ranibizumab therapy combined with TA versus ranibizumab monotherapy in patients with polypoidal choroidal vasculopathy (PCV). Furthermore, the pharmacogenetics effect of inflammatory related genes polymorphism in response to the treatments. To further confirm the role of inflammatory factors in the pathogenesis and advance of PCV.

DETAILED DESCRIPTION:
Polypoidal choroidal vasculopathy (PCV), a vascular disease of the choroid, appears to be the predominant subtype of exudative or "wet" AMD in Asian populations, in contrast to choroidal neovascularization secondary to AMD (CNV-AMD) in Western populations. There are distinct differences in pathophysiological, clinical and epidemiological factors between the two subtypes, although they also share some common risk factors. In contrast to CNV-AMD, PCV does not seem to respond as well to anti-VEGF treatment. The optimal treatment option for PCV remains elusive, with most studies showing good short-term visual outcome but poorer longer-term outcome with current treatment strategies. Therefore, understanding the pathogenesis of PCV, while developing novel and effective treatments strategies to prevent PCV-related vision loss is significant unmet needs.

The purpose of this study is to assess the effects and safety of ranibizumab therapy combined with TA versus ranibizumab monotherapy in patients with PCV. Second, the pharmacogenetics effect of inflammatory related genes and polymorphism in response to the treatments of PCV will be explored. To further confirm the role of inflammatory factors in the pathogenesis and advance of PCV, it is important to determine the levels of inflammatory factors in the anterior chamber aqueous humor from PCV patients, comparing with the aqueous humor acquired from the age-matched age-related cataract patients undergoing phacoemulsification.

ELIGIBILITY:
Inclusion Criteria:

* bestcorrected visual acuity (BCVA) letter score of 73 to 24 using Early Treatment of Diabetic Retinopathy Study charts at a starting distance of 4 m (20/40 to 20/320 Snellen equivalent);
* a greatest lineardimensionof the lesion of <5400 um( 9 Macular Photocoagulation Study disk areas), assessed by ICGA;
* Cross-reading by different center to conﬁrmed diagnosis of PCV, that is, presence of early subretinal focal ICGA hyperﬂuorescence (appearing within the ﬁrst 6 minutes after injection of indocyanine green) and in addition, at least one of the following angiographic or clinical criteria: (i) association with a BVN, (ii) presence of pulsatile polyp, (iii) nodular appearance when viewed stereoscopically, (iv) presence of hypoﬂuorescent halo (in ﬁrst 6 minutes),7 (v) orange subretinal nodules in stereoscopic color fundus photograph (polyp corresponding to ICGA lesions), or (vi) association with massive submacular hemorrhage (deﬁned as size of hemorrhage of at least 4 disk areas).

Exclusion Criteria:

* received treatment previously with verteporﬁn PDT, focal laser photocoagulation, transpupillary thermotherapy, pneumatic displacement of subretinal blood, or any investigational treatment;
* a history of angioid streaks, presumed ocular histoplasmosis syndrome, or pathologic myopia;
* experienced RPE tear, retinal detachment, macular hole, or uncontrolled glaucoma;
* undergone intraocular surgery (except uncomplicated cataract extraction with intraocular lens implantation within 60 days before the screening visit)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Change of mean BCVA | 12 months
  Change of Central BCVA (Measured with EDTRS Chart,numbers of letters) (primary: baseline and 6 months, secondary: baseline to 12 months)

SECONDARY OUTCOMES:
Change of Central Rerina Thickness | 12 months
  Change of Central Rerina Thickness (um) (primary: between baseline and 6 months, secondary: between baseline to 12 months)
regression of Branch vacular network(BVN) | 12 months
  Size of Branch vascular network (um)
Polyps regression | 12 months
  Size of polyps (um)(primary: between baseline and 6 months, secondary: between baseline to 12 months)
Number of re-treatments | 12 month
  re-treatments numbers

CONTACTS AND LOCATIONS:
Overall Officials: Shibo Tang, Study Chair — Aier School of Ophthalmology, Central South University
Locations (7):
- China (7):
  - Beijing Aier Intech Eye Hospital, Beijing, Beijing Municipality
  - Guangzhou Aier Eye Hospital, Guanzhou, Guangdong
  - Shenzhen Aier Eye Hospital, Shenzhen, Guangdong
  - Shenzhen Eye Hospital, Shenzhen, Guangdong
  - Harbin Aier Eye Hospital, Harbin, Heilongjiang
  - Wuhan General Hospital of PLA, Wuhan, Hubei
  - The Eye Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No